CLINICAL TRIAL: NCT03029260
Title: Effect of Nervous System Mobilization on Heat, Cold and Mechanical Pain Thresholds and Lower Limb Flexibility
Brief Title: Effects of Nervous System Mobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Dr, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NSM01
Record Dates: First submitted 2017-01-19; First posted 2017-01-24 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Healthy Individuals

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Neural mobilization - tension (Experimental): It is anticipated that 30 participants will be in this group. They will receive tension type neural mobilization of the peroneal nerve in the dominant limb. This will consist of positioning the lower limb with inversion and plantar flexion of the ankle, extension of the knee and maximum flexion of the hip without pain. A physiotherapists will move the hip from this maximum position of flexion in direction to extension (for example if the participants reaches 80º of flexion the mobilization will be between 40º and 80º of flexion). Each participant will receive four series of 10 mobilizations with 1 minute rest between series.
  Interventions: Other: Neural mobilization - tension.
- Neural mobilization - sliding (Active Comparator): It is anticipated that 30 participants will be in this group. They will receive sliding neural mobilization of the peroneal nerve in the dominant limb. Each participant will receive four series of 10 mobilizations with 1 minute rest between series of the following combination of movement: from ankle dorsiflexion, knee extension and hip extension to ankle plantarflexion, knee and hip flexion.
  Interventions: Other: Neural mobilization - gliding

INTERVENTIONS:
Other: Neural mobilization - tension. — Neural mobilization in tension consists of using combinations of joint movement known to maximize the tension and lengthening of peripheral nervous structures.
  The intervention will be delivered in one session only.
  Arms: Neural mobilization - tension
Other: Neural mobilization - gliding — Gliding neural mobilization consists of using combinations of joint movement known to maximize the movement of the peripheral nerves in relation to adjacent structures.
  The intervention will be delivered in one session only.
  Arms: Neural mobilization - sliding

SUMMARY:
This study aims to compare the effect of tension neural mobilization versus sliding neural mobilization of the peroneal nerve on the heat and cold threshold, on pressure pain threshold and on flexibility both in the dominant lower limb (subjected to mobilization) and the non-dominant lower limb (not subjected to mobilization) in healthy young participants.

DETAILED DESCRIPTION:
Sixty young and healthy participants will be randomly allocated to receive tension neural mobilization (n=30) or sliding neural mobilization (n=30). Data on heat threshold, cold threshold, pressure pain threshold and lower limb flexibility will be collected before the intervention, immediately after the intervention and at least 24h after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* naïve to nervous system mobilization;

Exclusion Criteria:

* Any surgery or trauma in the previous 6 months; neurological, cardiorespiratory or rheumatic pathology; cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Range of motion of the Straight Leg Raising test | Baseline
  The hip is raised to maximum flexion and the degree of flexion is measured with universal goniometer
Range of motion of the Straight Leg Raising test | Approximately 45 minutes after baseline measurements
  The hip is raised to maximum flexion and the degree of flexion is measured with universal goniometer
Range of motion of the Straight Leg Raising test | At least 24 hours after baseline measurements
  The hip is raised to maximum flexion and the degree of flexion is measured with universal goniometer

SECONDARY OUTCOMES:
Heat threshold | Baseline
  This is measured with a QSense instrument, which has thermode that is attached to the skin. The temperature in this thermode increases or decreases (as per the protocol being used) and the participants is holding a device to stop the temperature to increase/decrease when he/she first perceives it. The temperature perceived is the test result.
Heat threshold | Approximately 45 minutes after baseline measurements
  This is measured with a QSense instrument, which has thermode that is attached to the skin. The temperature in this thermode increases or decreases (as per the protocol being used) and the participants is holding a device to stop the temperature to increase/decrease when he/she first perceives it. The temperature perceived is the test result.
Heat threshold | At least 24 hours after baseline measurements
  This is measured with a QSense instrument, which has thermode that is attached to the skin. The temperature in this thermode increases or decreases (as per the protocol being used) and the participants is holding a device to stop the temperature to increase/decrease when he/she first perceives it. The temperature perceived is the test result.
Cold threshold | Baseline
  This is measured with a QSense instrument, which has thermode that is attached to the skin. The temperature in this thermode increases or decreases (as per the protocol being used) and the participants is holding a device to stop the temperature to increase/decrease when he/she first perceives it. The temperature perceived is the test result.
Cold threshold | Approximately 45 minutes after baseline measurements
  This is measured with a QSense instrument, which has thermode that is attached to the skin. The temperature in this thermode increases or decreases (as per the protocol being used) and the participants is holding a device to stop the temperature to increase/decrease when he/she first perceives it. The temperature perceived is the test result.
Cold threshold | At least 24 hours after baseline measurements
  This is measured with a QSense instrument, which has thermode that is attached to the skin. The temperature in this thermode increases or decreases (as per the protocol being used) and the participants is holding a device to stop the temperature to increase/decrease when he/she first perceives it. The temperature perceived is the test result.
Pressure pain threshold | Baseline
  This is measured using a pressure pain algometer. Pressure is made with this device against a specific body region (upper and lateral part of the dominant foot) until the participants perceives that the pressure changes to pain. The amount of pressure that the participants perceives as being painful is the test result.
Pressure pain threshold | Approximately 45 minutes after baseline measurements
  This is measured using a pressure pain algometer. Pressure is made with this device against a specific body region (upper and lateral part of the dominant foot) until the participants perceives that the pressure changes to pain. The amount of pressure that the participants perceives as being painful is the test result.
Pressure pain threshold | At least 24 hours after baseline measurements
  This is measured using a pressure pain algometer. Pressure is made with this device against a specific body region (upper and lateral part of the dominant foot) until the participants perceives that the pressure changes to pain. The amount of pressure that the participants perceives as being painful is the test result.

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Silva, PhD, Principal Investigator — University of aveiro
Locations (1):
- School of Health Sciences, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No